CLINICAL TRIAL: NCT00299234
Title: Atomoxetine for Children With Acquired Attentional Disorders Following Completion of Chemotherapy for Acute Lymphocytic Leukemia
Brief Title: Atomoxetine for Children With Acquired Attentional Disorders Following Completion of Chemotherapy for ALL
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient number of interested potentital subjects
Sponsor: Monarch Medical Research (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Donald W Lewis, MD, Children's Specialty Group
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B4Z-MC-X040
Record Dates: First submitted 2006-03-02; First posted 2006-03-06 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2007-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator): placebo
  Interventions: Drug: Atomoxetine
- 1 (Experimental): atomoxetine
  Interventions: Drug: Atomoxetine

INTERVENTIONS:
Drug: Atomoxetine — titration schedule: 0.5 to 1.5 mg/kg/day

SUMMARY:
This study is a double-blind, placebo-controlled, parallel group trial of atomoxetine (1.8 mg/kg) for the management of chemotherapy-related acquired attentional disorders in children who have survived Acute Lymphocytic Leukemia. Atomoxetine will produce a favorable impact on ADHD symptoms in children with chemo-related acquired attentional disorders.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the safety, tolerability and efficacy of atomoxetine as determined by the change in the ADHD-RS-IV Total score compared to placebo in the symptomatic treatment of patients diagnosed with Attention-Deficit/Hyperactivity Disorder (by DSM-IV ADHD-NOS criteria) occurring as a neuropsychological late-effect of chemotherapy used to treat Acute Lymphocytic Leukemia (ALL).

The secondary objectives are:

1. to assess the effect of once daily (AM) dosing of atomoxetine (1.8mg/kg) compared to placebo on ADHD symptoms as measured by:

   * ADHD-RS Total score inclusive of subtypes for inattention, hyperactivity and combined subtypes.
   * Clinical Global Impression-ADHD
2. to evaluate the safety and tolerability of atomoxetine compared with placebo based on treatment-emergent adverse events (AEs), laboratory tests, vital signs, physical examinations, and ECGs.

ELIGIBILITY:
Inclusion Criteria:

* Ages 6-18 years
* Must have successfully completed treatment for ALL and are currently 1-year "disease free" as judged by the investigators.
* Must meet DSM-IV criteria for "ADHD-NOS.( Attachment A) The attention deficit symptoms have been precipitated by chemotherapy-related neurological injury. Therefore, the DSM-IV category is ADHD-NOS.
* Must have an Investigator-completed ADHD-RS total and/or subscale score of ≥1.5 standard deviations above age/gender norm.
* Laboratory results, including chemistries, hematology, and urinalysis do not demonstrate clinically significant abnormalities.
* ECG demonstrates no clinically significant abnormalities
* Educational level and degree of understanding of the patient and their parents permit suitable communication between the investigators and study coordinators.
* Subjects and parents are judged to be reliable to keep appointments.
* Must be able to swallow tablets.
* Must have demonstrated compliance during their chemotherapy program.
* Must weigh > 20 kg.

Exclusion Criteria:

* Have relapsed or are having re-occurring symptoms/signs of ALL.
* Have had substantial exposure to radiation therapy (>2000: cGy) since high dose radiation treatment is associated with neurocognitive deficits or be "treatment resistant" pharmacologically.
* Past exposure to atomoxetine.
* ADHD symptoms or treatment prior to the diagnosis of ALL
* Documented bipolar disorder, psychosis, affective disorder.
* Female subjects who are pregnant or breastfeeding.
* Suicide risk.
* Seizure disorders (except history of febrile seizures).
* Histories of multiple drug allergies.
* Histories of alcohol or substance abuse.
* Prior or current medical conditions that, in the opinion of the investigators, could be exacerbated by atomoxetine.
* Sympathomimetic overactivity such as catecholamine secreting tumor.
* Use of MAOI medications.
* Have taken psychostimulants one week prior to randomization.
* Current or past history of hypertension.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2006-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the change in the ADHD-RS total score from baseline to completion of the study. | 5 weeks

SECONDARY OUTCOMES:
The secondary outcome is the difference in CGI categories by the treatment versus placebo group. | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Donald W Lewis, MD, Principal Investigator — Monarch Medical Research
Locations (1):
- Monarch Medical Research - Child and Adolescent Neurology, Norfolk, Virginia, United States

REFERENCES:
- [Background] Mulhern RK, Friedman AG, Stone PA. Acute lymphoblastic leukemia: long-term psychological outcome. Biomed Pharmacother. 1988;42(4):243-6. PMID 3056531
- [Background] Schuler D, Bakos M, Borsi J, Gacsaly I, Kalmanchey R, Kardos G, Koos R, Nagy C, Revesz T, Somlo P, et al. Neuropsychologic and CT examinations in leukemic patients surviving 10 or more years. Med Pediatr Oncol. 1990;18(2):123-5. doi: 10.1002/mpo.2950180207. PMID 2304419
- [Background] Goff JR, Anderson HR Jr, Cooper PF. Distractibility and memory deficits in long-term survivors of acute lymphoblastic leukemia. J Dev Behav Pediatr. 1980 Dec;1(4):158-63. PMID 6941969